CLINICAL TRIAL: NCT05567523
Title: Effects of Dexmedetomidine at Different Doses on Hemodynamics and Recovery Quality in Elderly Patients Undergoing Hip Replacement Surgery Under General Anesthesia
Brief Title: Safety Study of Dexmedetomidine in Elderly Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhenjiang First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SQK-20190131-W
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hip Fractures; Hip Disease
Keywords: Dexmedetomidine; Elderly; Hemodynamics; Hip replacement; General anesthesia
MeSH Terms: conditions — Hip Fractures | interventions — Dexmedetomidine; Saline Solution; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D0.25, Group D0.5, Group D0.75 (Experimental): Dexmedetomidine will be administered at different initial loading doses (0.25/0.5/0.75 μg/kg within 15min) following same maintained dosage ( 0.5μg/kg/h) in Group D0.25/D0.5/D0.75.
  Interventions: Drug: Dexmedetomidine
- Group NS, Group MD (Placebo Comparator): In Group NS, patients will be pumped 0.1ml/kg of normal saline for 15min before anesthesia induction, following continuous infusion at the rate of 0.125ml/kg/h until the end of operation. In Group MD, patients will be administrated with midazolam 0.03mg/kg at the beginning of anesthesia induction.
  Interventions: Drug: Normal saline; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — In dexmedetomidine groups, patients will be pumped 0.1ml/kg of dexmedetomidine (contained dexmedetomidine 0.25/0.5/0.75µg/kg in Group D0.25/D0.5/D0.75) for 15min before anesthesia induction, following continuous infusion at the rate of 0.125ml/kg/h until the end of operation.
  Other Names: Dex
  Arms: Group D0.25, Group D0.5, Group D0.75
Drug: Normal saline — normal saline
  Other Names: physiological saline
  Arms: Group NS, Group MD
Drug: Midazolam — midazolam
  Other Names: Dormicum
  Arms: Group NS, Group MD

SUMMARY:
The purpose of this study is to find out appropriate dose range of dexmedetomidine to provide the elderly patients satisfactory sedation and analgesia with stable hemodynamics during perioperative period of hip replacement under general anesthesia.

DETAILED DESCRIPTION:
All patients will be screened to determine eligibility for study entry, and the patients who meet the eligibility requirements will be informed about the study and potential risks. After giving written informed consent, the patients will be randomized into different doses of dexmedetomidine groups and the comparative groups in a same ratio.

ELIGIBILITY:
Inclusion Criteria:

* age ≥65yr, American Society of Anesthesiologists (ASA) physical status scale grade I-III, ready for HP; body weight between 45 and 75kg, body mass index (BMI) between 18 and 24kg/m2;
* the health conditions generally well according to medical history, physical examination, and laboratory tests;
* no signs of difficult intubation;
* no history of dementia and mental problems;
* normal cognitive function, ability to understand and comply with study procedures.

Exclusion Criteria:

* Age <65 yr or >90 yr; BMI greater than 24 kg/m2; ASA grade higher than III;
* Heart failure, severe arrhythmias, severe bradycardia (heart rate less than 40 beats/min), atrioventricular block of degree 2 or above, sick sinus syndrome, systolic blood pressure (SBP) ≥180 or <90 mmHg, diastolic blood pressure (DBP) ≥110 or <60 mmHg;
* Severe liver or kidney dysfunction, severe infection, and other pathological conditions that interfere with study results.
* Dementia, cerebrovascular accidents within 3 months, mental illness, epilepsy, and other adverse events that interfere with study results.
* Patients with the conditions that block communication and preoperative assessment, such as serious hearing or visual impairment;
* History of chronic analgesic use, long-term psychotropic medication use, alcohol or drug addiction.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Changes of baseline blood pressure | Through the whole perioperative period, an average of 10 hours
  Changes of baseline blood pressure in each group, including systolic blood pressure, diastolic blood pressure and mean arterial pressure
Changes of baseline heart rate | Through the whole perioperative period, an average of 10 hours
  Changes of baseline heart rate in each group
Numbers of elderly patients with hypotension | Through the whole perioperative period, an average of 10 hours
  Hypotension is defined as systolic blood pressure <90 mmHg or mean arterial pressure below >20% of basal values.
Numbers of elderly patients with bradycardia | Through the whole perioperative period, an average of 10 hours
  Bradycardia is defined as heart rate <50 beats/min or below >20% of basal values.

SECONDARY OUTCOMES:
Sedation changes after general anesthesia using Richmond agitation-sedation scale | before general anesthesia, up to 2 hours after general anesthesia
  Sedation changes after general anesthesia using Richmond agitation-sedation scale(-5 to +4, 0 means awake and quiet) in each group
Pain changes after general anesthesia using visual analogue scale | before general anesthesia, up to 2 hours after general anesthesia
  Pain changes after general anesthesia using visual analogue scale(0 to 10,higher scores mean a worse outcome) in each group

CONTACTS AND LOCATIONS:
Overall Officials: Haitong Liu, Study Director — Zhenjiang First People's Hospital
Locations (1):
- Zhenjiang First People's Hospital, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Data are available after publication and up to one year after publication.
Access Criteria: Send an email to dolinet@163.com

REFERENCES:
- [Background] Colin PJ, Hannivoort LN, Eleveld DJ, Reyntjens KMEM, Absalom AR, Vereecke HEM, Struys MMRF. Dexmedetomidine pharmacokinetic-pharmacodynamic modelling in healthy volunteers: 1. Influence of arousal on bispectral index and sedation. Br J Anaesth. 2017 Aug 1;119(2):200-210. doi: 10.1093/bja/aex085. PMID 28854538
- [Background] Colin PJ, Hannivoort LN, Eleveld DJ, Reyntjens KMEM, Absalom AR, Vereecke HEM, Struys MMRF. Dexmedetomidine pharmacodynamics in healthy volunteers: 2. Haemodynamic profile. Br J Anaesth. 2017 Aug 1;119(2):211-220. doi: 10.1093/bja/aex086. PMID 28854543
- [Background] Le Bot A, Michelet D, Hilly J, Maesani M, Dilly MP, Brasher C, Mantz J, Dahmani S. Efficacy of intraoperative dexmedetomidine compared with placebo for surgery in adults: a meta-analysis of published studies. Minerva Anestesiol. 2015 Oct;81(10):1105-17. Epub 2015 May 25. PMID 26005187
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Liu Y, Ma L, Gao M, Guo W, Ma Y. Dexmedetomidine reduces postoperative delirium after joint replacement in elderly patients with mild cognitive impairment. Aging Clin Exp Res. 2016 Aug;28(4):729-36. doi: 10.1007/s40520-015-0492-3. Epub 2015 Nov 11. PMID 26559412
- [Background] Mei B, Meng G, Xu G, Cheng X, Chen S, Zhang Y, Zhang M, Liu X, Gu E. Intraoperative Sedation With Dexmedetomidine is Superior to Propofol for Elderly Patients Undergoing Hip Arthroplasty: A Prospective Randomized Controlled Study. Clin J Pain. 2018 Sep;34(9):811-817. doi: 10.1097/AJP.0000000000000605. PMID 29528863
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Wang BJ, Li CJ, Hu J, Li HJ, Guo C, Wang ZH, Zhang QC, Mu DL, Wang DX. Impact of dexmedetomidine infusion during general anaesthesia on incidence of postoperative delirium in elderly patients after major non-cardiac surgery: study protocol of a randomised, double-blinded and placebo-controlled trial. BMJ Open. 2018 Apr 21;8(4):e019549. doi: 10.1136/bmjopen-2017-019549. PMID 29680809
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Kim SY, Kim JM, Lee JH, Song BM, Koo BN. Efficacy of intraoperative dexmedetomidine infusion on emergence agitation and quality of recovery after nasal surgery. Br J Anaesth. 2013 Aug;111(2):222-8. doi: 10.1093/bja/aet056. Epub 2013 Mar 22. PMID 23524149
- [Derived] Liu H, Gao M, Zheng Y, Sun C, Lu Q, Shao D. Effects of dexmedetomidine at different dosages on perioperative haemodynamics and postoperative recovery quality in elderly patients undergoing hip replacement surgery under general anaesthesia: a randomized controlled trial. Trials. 2023 Jun 8;24(1):386. doi: 10.1186/s13063-023-07384-z. PMID 37291651